CLINICAL TRIAL: NCT06447272
Title: Effects of Inspiratory Muscle Training on Respiratory and Diaphragmatic Functions, Balance Control, Exercise Capacity and Quality of Life in People After Stroke: a Randomized Controlled Trial
Brief Title: Effects of IMT on Respiratory, Diaphragmatic and Balance Functions, Exercise Capacity and QOL in People After Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, LIU FANG, Principal Investigator, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE-OT2023/13
Record Dates: First submitted 2024-05-28; First posted 2024-06-07 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Stroke; Inspiratory muscle training; Diaphragm; Balance control; Exercise capacity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham IMT (Sham Comparator): conventional treatment + sham IMT
  Interventions: Other: sham inspiratory muscle training
- Target IMT (Experimental): conventional treatment + target IMT
  Interventions: Other: target inspiratory muscle training

INTERVENTIONS:
Other: sham inspiratory muscle training — This group will receive conventional treatment + sham IMT (with 10% MIP as the training intensity)
  Arms: Sham IMT
Other: target inspiratory muscle training — This group will receive conventional treatment + target IMT (the IMT identified as optimal intensity based on the results of our undergoing study).
  Arms: Target IMT

SUMMARY:
This is a randomized controlled trial. This current RCT study will be a continuing project based on the optimal IMT intensity identified from our ongoing study. This ongoing study (registered on ClinicalTrials.gov with the registration number NCT06267768) aims to explore the optimal IMT intensity for the recruitment of diaphragm muscles in people after a stroke. Based on this intensity, the aim of this RCT is to explore the effects of a 4-week protocol of IMT on respiratory function, balance control, exercise capacity, and quality of life in people after a stroke.

ELIGIBILITY:
Inclusion Criteria:

* aged between 40 and 80 years;
* breathing spontaneously;
* clinically diagnosed with ischemic and/or haemorrhagic stroke;
* stroke duration from onset between 1 and 12 months;
* no history of thoracic or abdominal surgery within the last 6 months;
* able to understand and follow verbal instructions;
* no facial palsy, or mild facial palsy without limitation of labial occlusion;
* capable of maintaining a resting sitting posture without feet support for at least 30 seconds;
* no cognitive impairment, as indicated by a Montreal Cognitive Assessment (MoCA) score of ≥ 26;
* able to independently walk at least 10 meters with or without an assistive device.

Exclusion criteria:

* acute myocardial infarction or acute heart failure;
* acute pain in any part of the body;
* with respiratory illness or positive clinical signs of impaired respiratory function, such as shortness of breath, hypoxemia, chronic cough, or sputum retention;
* with chronic cardiovascular dysfunction;
* Trunk Impairment Scale (TIS) score ≥ 20;
* presence of a nasal feeding tube, tracheal tube, or any condition that prevents the measurement or implementation of the study procedure.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic thickness | baseline, after 4 weeks of intervention
  The diaphragmatic thickness of both the left and right diaphragms will be measured by ultrasound. (Mindray M9, Shenzhen, China).

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | baseline, after 4 weeks of intervention
  Forced Vital Capacity (FVC) is a measurement used in pulmonary function tests to assess lung function. It refers to the total volume of air that a person can forcibly exhale from their lungs after taking the deepest breath possible. It will be measured using the spirometer.
Forced Expiratory Volume in one second (FEV1) | baseline, after 4 weeks of intervention
  Forced Expiratory Volume in one second (FEV1) measures the volume of air a person can forcibly exhale in the first second of a forced breath. It will be measured using the spirometer.
Maximum Inspiratory Pressure (MIP) | baseline, after 4 weeks of intervention
  Maximum Inspiratory Pressure (MIP) is a measure used in pulmonary function testing to assess the strength of the respiratory muscles, particularly the muscles used for inhalation. It will be measured using the spirometer.
Trunk Impairment Scale (TIS) | baseline, after 4 weeks of intervention
  The TIS is a rating scale used to measure static sitting balance, dynamic sitting balance, and trunk coordination. The total TIS score ranges from 0 to 23 points, with a higher score indicating better trunk function.
Sitting Balance | baseline, after 4 weeks of intervention
  A force plate will be used to measure changes in the center of pressure during the performance of various tasks in sitting positions.
Timed Up and Go Test (TUG) | baseline, after 4 weeks of intervention
  TUG is a test to measure the time that a participant needs to stand up from a standard armchair, walk a short distance of about 3 meters, turn around, walk back to the chair, and sit down again.
Falls efficacy scale international | baseline, after 4 weeks of intervention, 12-week follow-up after the end of intervention
  The Falls Efficacy Scale-International (FES-I) is a questionnaire measuring fear of falling in older adults. It consists of 16 items, each scored from 1 to 4, with higher scores indicating greater fear. The total score ranges from 16 (lowest fear) to 64 (highest fear). It is used in clinical settings to assess fall risk and tailor interventions.
6-Minute Walk Test | baseline, after 4 weeks of intervention
  The 6-Minute Walk Test (6MWT) measures how far someone can walk in six minutes. It assesses exercise capacity and mobility.
Stroke Impact Scale | baseline, after 4 weeks of intervention, 12-week follow-up after the end of intervention
  The Chinese version of the Stroke Impact Scale 3.0 (SIS) will be used to measure the quality of life. Scores range from 0 to 100, a higher overall score suggests better physical, emotional, and social functioning, while a lower score may indicate more significant impairment or limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Fang LIU, Principal Investigator — Hong Kong Metropolitan University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT06447272/Prot_SAP_004.pdf
  • Informed Consent Form (2025-01-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT06447272/ICF_005.pdf